CLINICAL TRIAL: NCT01011972
Title: A Phase 1 Study of the Safety and Pharmacokinetics of XMT-1107 Administered as an Intravenous Infusion Once Every Three Weeks to Patients With Advanced Solid Tumors
Brief Title: A Study of Intravenous XMT-1107 in Patients With Advanced Solid Tumors
Acronym: XMT-1107
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mersana Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MER-1107-001
Record Dates: First submitted 2009-11-10; First posted 2009-11-11 (Estimated); Last update posted 2018-01-31 (Actual); Status verified 2016-09

CONDITIONS: Neoplasm Metastasis
Keywords: Dose escalation; XMT-1107; 1107; Tumor; Phase 1; Fumagillol; PHF; Fleximer; cancer; maximum tolerated dose; MTD
MeSH Terms: conditions — Neoplasm Metastasis; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- XMT-1107 (Experimental): Dose escalation groups of XMT-1107, I.V. (in the arm) beginning at 6 mg/m^2, doubling in dose to 24 mg/m^2, then 40 mg/m^2, then 60 mg/m^2, then 80 mg/m^2 with subsequent doses at 33% of the previous until disease progression or unacceptable side effects are experienced.
  Interventions: Drug: XMT-1107

INTERVENTIONS:
Drug: XMT-1107 — 6 mg XMT-1107 administered by I.V. (in the vein) administered over 90 min, once every 21 days : until progression or unacceptable toxicity develops
  Other Names: conjugated XMT-1191

SUMMARY:
XMT-1107 has been shown in nonclinical studies to slow the growth of tumors. These effects may result from blocking the growth of new blood vessels that help the tumors survive.

DETAILED DESCRIPTION:
This is an open-label, ascending-dose study of XMT-1107 administered intravenously over 90 minutes every 21 days (1 cycle). Blood sampling for PK analyses will be performed immediately prior to dosing and after dosing. Adverse events will be graded according to the National Cancer Institute (NCI) Common Terminology Criteria (CTC) version 4.0 (CTCAE v4.0)

ELIGIBILITY:
Inclusion Criteria:

* Patient must have a histological diagnosis of advanced solid tumor and must be refractory to standard therapy or have no effective therapy.
* Measurable or evaluable disease.
* At least 42 days since administration of mitomycin or nitrosoureas and 28 days since any other chemotherapy, investigational agent, and/or radiation therapy.
* Age ≥ 18 years old.
* Have the following laboratory values:

  * Absolute neutrophil count (ANC) ≥ 1500 cells/mm3
  * Platelet count ≥ 100,000 cells/mm3
  * Hemoglobin ≥ 9 g/dL
  * Serum creatinine ≤ 1.5 mg/dL or calculated creatinine clearance ≥ 60 mL/min (Calculated by Cockroft and Gault method. Creatinine clearance (mL/min) = (140-age) x weight (kg)/72 x (serum creatinine in mg/dL) = ml**/min (**for females, multiply results by 0.85))
  * Total bilirubin ≤ 1.5 mg/dL or ≤ upper limit of normal (ULN)
  * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 times the institutional upper limit of normal (ULN) or ≤ 5 times ULN of liver metastases are present
  * Prothrombin time (PT) and partial thromboplastin time (PTT) ≤ 1.5 times the ULN
* Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) 0-1.
* Life expectancy of at least 3 months.
* Signed informed written consent.

Exclusion Criteria:

* Known brain metastases (either currently or previously).
* Peripheral neuropathy ≥ Grade 2.
* Ataxia ≥ Grade 1.
* Cognitive disturbance ≥ Grade 1.
* History of seizures.
* Patients known to be human immunodeficiency virus (HIV) positive.
* Active infections requiring IV antibiotics or serious intercurrent illness, including hepatitis B or C.
* Unstable angina, recent myocardial infarction (within the previous 6 months), or use of ongoing maintenance therapy for life-threatening arrhythmia.
* Known hypersensitivity to this class of drugs.
* Pregnant or nursing women, women who are of childbearing potential and are not using an effective method of either barrier or hormonal contraceptives. Men who are not using an effective method of barrier contraceptive, or who would not be willing to continue to use these effective methods for the duration of the study.
* Patients who have had a major surgical procedure (not including mediastinoscopy), open biopsy, or significant traumatic injury ≤ 4 weeks prior to beginning treatment.
* Patients with proteinuria at screening as demonstrated by either:

  1. urine protein creatinine (UPC) ratio ≥ 1.0 at screening OR
  2. urine dipstick for proteinuria ≥ 2+ (patients discovered to have ≥ 2+ proteinuria on dipstick urinalysis at baseline should undergo a 24 hour urine collection, and must demonstrate ≤ 1 g of protein/24 hours to be eligible)
* Patients with a serious non-healing wound, active ulcer, or untreated bone fracture.
* Patients with history of hematemesis or hemoptysis (defined as having bright red blood of ½ teaspoon or more per episode) ≤ 1 month prior to study enrollment.
* Inadequately controlled hypertension (defined as systolic blood pressure >140 mm Hg and/or diastolic blood pressure > 90 mm Hg while on antihypertensive medications). Initiation of antihypertensive agents is permitted provided adequate control is documented at least 1 week prior to beginning study treatment.
* Significant vascular disease (e.g., aortic aneurysm requiring surgical repair, or recent peripheral arterial thrombosis) ≤ 6 months prior to Day 1 of treatment.
* History of stroke or transient ischemic attack ≤ 6 months prior to beginning treatment.
* Any prior history of hypertensive crisis or hypertensive encephalopathy.
* History of abdominal fistula or gastrointestinal perforation ≤ 6 months prior to Day 1 of beginning treatment.
* QTc interval > 470 milliseconds as calculated by Bazett's formula.
* Any issue that, in the opinion of the Investigator, would render the patient unsuitable for study participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2010-03 (Actual); Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
The primary objective of this study is to determine the maximum tolerated dose of XMT-1107 when given via IV once every three weeks. | Adverse events are assessed during each treatment cycle.

SECONDARY OUTCOMES:
Assess the pharmacokinetics (PK) of XMT-1107 and its release product | Samples for PK are collected during Cycle 1 and prior to each subsequent treatment cycle
Determine the recommended Phase 2 dose of XMT-1107 | Throughout Cycle 1
Assess the safety of XMT-1107. | Throughout Cycle 1
Observe for evidence of anti-tumor activity by XMT-1107. | Course of study
Monitor the effect of XMT-1107 on MetAP2 inhibition in leukocytes from patients | Cycle 1 and Cycle 2

CONTACTS AND LOCATIONS:
Overall Officials: Johana Bendell, MD, Principal Investigator — Sara Cannon Research Institute; Geoffrey Shapiro, MD, Principal Investigator — Dana-Farber Cancer Institute; Edward Sausville, MD, Principal Investigator — University of Maryland, Greenbaum Cancer Center
Locations (4):
- United States (4):
  - University of MD Greenbaum Cancer Center, Baltimore, Maryland
  - Dana Farber Cancer Institute (DFCI), Boston, Massachusetts
  - Beth Israel Deaconess Medical Center (BIDMC), Boston, Massachusetts
  - Sarah Cannon Research Institute (SCRI), Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No